CLINICAL TRIAL: NCT03919981
Title: A European, Multicenter, Prospective Clinical Study to Evaluate Cysteamine Toxicity on Human Osteoclasts. The CYSTEA-BONE Clinical Study.
Brief Title: CYSTEA-BONE Clinical Study
Acronym: CYSTEA-BONE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0685; 2019-A00166-51 (Other: ID-RCB)
Record Dates: First submitted 2019-02-21; First posted 2019-04-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Nephropathic Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 25 mL blood sample will be collected on citrate tubes for osteoclastic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nephropathic cystinosis patients receiving cysteamine: nephropathic cystinosis patients receiving cysteamine. The blood samples of the group will be used to evaluate the action of cysteamine on osteoclastic differentiation and resorption activity of NC patients, depending on the underlying genotype.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 25 mL blood sample will be collected on citrate tubes for osteoclastic analysis.

SUMMARY:
Nephropathic Cystinosis (NC) is an orphan inherited autosomal recessive disease characterised as a generalized lysosomal storage disease due to a deficiency of the cystine lysosomal transport protein, cystinosin.

Patients with NC usually receive cysteamine. Bone impairment was recently recognized as a late complication of NC, occurring at adolescence or early adulthood. Even though the exact underlying pathophysiology is unclear, at least six hypotheses are discussed, and mainly cysteamine toxicity and/or direct bone effect of the Cystinosin (CTNS) mutation. Because of the potential dramatic impact on quality of life of this novel complication, research should aim to better understand bone disease in NC.

The primary objective of this study is to evaluate the action of cysteamine on osteoclastic differentiation and resorption activity of NC patients, depending on the underlying genotype. The Secondary objective is to describe the clinical bone status of NC patients depending on their underlying genotype.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with confirmed diagnosis of nephropathic cystinosis (defined by clinical signs, White Blood Cells (WBC) cystine level and/or mutation), currently receiving oral cysteamine.
* Age > 2 years.
* Subjects and/or their parents/ legal guardian must provide non opposition prior to participation in the study.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nephropathic cystinosis (NC)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of positive Tartrate-resistant acid phosphatase (TRAP) cells | 1 day
  Number of positive TRAP cells will be assessed at the end of osteoclast differentiation from circulating monocytes

CONTACTS AND LOCATIONS:
Locations (13):
- France (10):
  - CHU de Besançon, Besançon
  - CHU Bordeaux - Hôpital Pellegrin tripode, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Jeanne de Flandre, Lille
  - Hopital Edouard Herriot, Lyon
  - AP-HM - Timone Enfants, Marseille
  - CHU Paris - Hôpital Robert Debré, Paris
  - CHU Paris - Hôpital Necker-Enfants Malades, Paris
  - Hôpital des Enfants, Toulouse
  - CHRU Nancy - Hôpital Brabois Enfants, Vandœuvre-lès-Nancy
- Klinik für Pädiatrische Nieren-, Leber- und Stoffwechselerkrankungen, Hanover, Germany
- IRCCS Ospedale Pediatrico Bambino Gesù, Roma, Italy
- Hacettepe University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No